CLINICAL TRIAL: NCT03334591
Title: Research On the Optimized Treatment Method For Apatinib's Cure Of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYF001
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Two Different Treatment Methods
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib 5 days' continuous use and 2 days' off (Experimental): Apatinib 500mg 5 days' continuous use and 2 days' off with Docetaxel60mg/m2 to treat advanced gastric cancer
  Interventions: Drug: Apatinib
- Apatinib 500mg continuous use (Active Comparator): Apatinib 500mg continuous use with Docetaxel60mg/m2 to treat advanced gastric cancer
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg with Docetaxel 60mg/m2

SUMMARY:
The investigators hope that after this research, two different treatment methods' curative effects for advanced gastric cancer can be assessed. One is continuous use of apatinib, the other is 5 days' continuous use and 2 days' off of apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients,age≥18years
2. Confirmed by Pathology or histology of Gastric cancer
3. Patients who failed first-line chemotherapy
4. The ECOG physical status score:0 to 2
5. Expected survival ≥3months
6. Patients should be voluntary to the trail and provide with signed informed consent.
7. The researchers believe patients can benefit from the study.

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with a knowm history of allergic reactions and/ou hypersensitivity attributed to apatinib or its accessories
3. Patients with apatinib contraindications
4. Patients of doctors considered unsuitable for the trail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
progress free survival(PFS) | 1 year
  From data of randomization until the date of first dccumentde progression or date of death from any cause

SECONDARY OUTCOMES:
disease control rate (DCR) | 1year
  investigators will assess treatment response according to Response Evaluation Criteria in Soid Tumor
Objective tumor response rate(ORR) | 1year
  difined as the percentage of subjects having achieved confirmed Complete Response+Partial Response as best overall response according to radiological assessments
overall survival (os) | 1year
  difined as the length of time from random assignment to death or to last contact
Quality of life score | 1 year
  a questionnaire developed to assess the quality of life of cancer patients
adverse events | 1 year
  adverse events are evaluated according to National Cancer institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: yifu He, doctor, Study Chair — Anhui Provincial Cancer Hospital
Locations (1):
- Anhui Provincial Cancer Hospital, Hefei, Anhui, China

REFERENCES:
- [Derived] Yan Y, Li H, Wu S, Wang G, Luo H, Niu J, Cao L, Hu X, Xu H, Jia W, Sun Y, Yao Y, Chen W, Ke L, Hu B, Ji C, Sun Y, Chen J, Li M, He Y. Efficacy and safety of intermittent versus continuous dose apatinib plus docetaxel as second-line therapy in patients with advanced gastric cancer or gastroesophageal junction adenocarcinoma: a randomized controlled study. Ann Transl Med. 2022 Feb;10(4):205. doi: 10.21037/atm-22-546. PMID 35280426